CLINICAL TRIAL: NCT00951782
Title: Deep High-Frequency Repetitive Transcranial Magnetic Stimulation for Smoking Cessation in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Deep High-Frequency Repetitive Transcranial Magnetic Stimulation for Smoking Cessation
Acronym: TMS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BeerYaakov Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Pinhas Dannon, Prof. Pinhas Dannon, BeerYaakov Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 234-CTIL
Record Dates: First submitted 2009-07-14; First posted 2009-08-04 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Smoking
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- High frequency TMS + smoking cue (Active Comparator)
  Interventions: Device: High frequency TMS
- Sham TMS + smoking cue (Sham Comparator)
  Interventions: Device: Sham TMS
- Low frequency TMS +smoking cue (Active Comparator)
  Interventions: Device: Low frequency TMS
- Sham TMS - no cue (Sham Comparator)
  Interventions: Device: Sham TMS
- High frequency TMS - no cue (Active Comparator)
  Interventions: Device: High frequency TMS
- Low frequency - no cue (Active Comparator)
  Interventions: Device: Low frequency TMS

INTERVENTIONS:
Device: High frequency TMS — deep TMS HADD coil
  Arms: High frequency TMS + smoking cue; High frequency TMS - no cue
Device: Sham TMS — sham deep TMS HADD coil
  Arms: Sham TMS + smoking cue; Sham TMS - no cue
Device: Low frequency TMS — Deep TMS - HADD coil
  Arms: Low frequency - no cue; Low frequency TMS +smoking cue

SUMMARY:
Deep transcranial magnetic stimulation (TMS) is currently being evaluated as a treatment option in major depression. It has been shown to be a safe procedure . Deep transcranial magnetic stimulation coils are designed to maximize the electrical field deep in the brain by the summation of separate fields projected into the skull from several points around its periphery. The device is planned to minimize the accumulation of electrical charge on the surface of the brain. Such accumulation can give rise to an electrostatic field that might reduce the magnitude of the induced electric field both at the surface and inside, thus reducing the depth penetration of the induced electric field . Deep transcranial magnetic stimulation could be more effective than repetitive transcranial magnetic stimulation due to its deeper penetration into brain tissues . The deeper penetration should produce greater action on nerve fibers connecting the prefrontal cortex to the limbic system.

The ability of high-frequency repetitive transcranial magnetic stimulation (rTMS) to alter dopaminergic neurotransmission in subcortical structures could explain recent reports, which suggest that it has the potential to reduce smoking and nicotine craving. Ecihhammer et al demonstrated a reduction in the number of cigarettes smoked and in the desire to smoke after a single rTMS treatment (Eichhammer et al., 2003). In addition, Johan et al in a cross-over, double-blind, placebo-controlled study demonstrated a reduction in cigarette consumption and desire to smoke after a single repetitive transcranial magnetic stimulation treatment (Johann et al., 2003). Recently, the investigators have finished a complete study on nicotine addiction using repetitive transcranial magnetic stimulation for 10 consecutive days. They have found that 10 days of rTMS reduced significantly better from placebo the number of cigarettes smoked, nicotine dependence and craving (Amiaz et al 2007, in preparation). Interestingly, some of the effects were stronger in the sub-group of patients that were presented with smoking-related pictures immediately prior to stimulation onset. Although, these results are interesting and exciting, they have two important caveats. First, only about 50%-60% of the smokers responded to the repetitive transcranial magnetic stimulation treatment. Second, among those responded to the treatment, only 10% had quit totally from smoking. Therefore, the potential therapeutic benefit of this treatment is limited. The investigators' hypothesis is that deep transcranial magnetic stimulation may be more efficient in smoking cessation due to it's deeper penetration and therefore it's capability to stimulate deeper fibers of the dopamine-reward-activating system.

DETAILED DESCRIPTION:
Research Plan

I. PARTICIPANTS Male and female cigarette smokers who suffer from COPD. From the general population aged 21-70 who wishes to quit smoking and failed to respond to previous anti-smoking treatment. They will be recruited by advertisements in the newspapers and specific websites. The number of participants in each sub-group (as described in the table below) will be 15-17. The investigators will recruit 90-102 subjects over two years.

II. SCREENING PROCEDURE

Before stimulation procedures onset, participants will undergo a clinical interview. All subject candidates will give written informed consent to take part in the study. Thereafter, they will be tested for their baseline pretreatment level of nicotine addiction in a screening meeting. This includes a report on the level of consumption (number of cigarettes smoked per day and overall duration in years) and a visual analog scale (VAS, see below for details). In addition, a urine sample for cotinine levels (nicotine metabolite) will be obtained in order to objectively measure levels of nicotine. In addition, several self-administered questionnaires will be given to the subjects in order to measure their baseline craving and nicotine dependence:

1. Fagerstrom Test of Nicotine Dependence (FTND) (Heatherton et al., 1991). (Appendix no.1a)
2. Tobacco Craving Questionnaire (TCQ) (Heishman et al., 2003). (Appendix no.1b)
3. Full demographic questionnaire about medical condition and smoking habits. (Appendix no.1c)

III. MEASURES

All subjects will undergo various measurements on several visits, as described in table 1-3, for nicotine consumption, craving and dependence during the rTMS treatment visits:

1. VAS: Visual Analogue Scale, on which the subject marks his/her subjective craving on a 10-cm-long scale in response to the following question: "How much do you crave a joint/bong right now?" This "desire to smoke rating" has been shown to be sensitive to assess self-reported levels of craving in nicotine smoking (Schuh and Stitzer, 1995; King and Meyer, 2000).
2. Short TCQ: Tobacco Craving Questionnaire, the short version of the TCQ, which has 12 questions that can be divided into four categories: emotionality, expectancy, compulsivity and purposefulness.
3. FTND: Fagerstrom Test of Nicotine Dependence. Measures the level of nicotine dependence (Dijkstra and Tromp, 2002).
4. Self-report of the number of cigarettes smoked on the previous day.
5. Urine sample.
6. BR: desire to smoke and effect on hunger.
7. Spatial span memory test - in order to evaluate the effect of deep rTMS on spatial memory. This test will be conducted in the screening interview and after 10 days of rTMS treatment.

IV. PRESENTATION OF PHOTOGRAPHS

It has recently been demonstrated that in nicotine-deprived smokers, reward and attention circuits are reactivated by mere exposure to smoking-related images, in contrast with neutral images (Due et al., 2002). In our experiment, prior to stimulation onset 14 'neutral' or 'nicotine-related' colored photographs will be presented on a computer screen to the participants while there are seated. The 'nicotine-related' photographs will be composed from smoking-related scenes, such as lighting up a cigarette, smoking puffs etc. 'Neutral' photos will consist of matched pictures without any nicotine related content (e.g. inanimate objects, hands, faces etc.). As the investigators have previously shown with the figure-8 coil experiment, there was a stronger effect of the rTMS treatment in subjects exposed to the nicotine photographs. The investigators propose that presentation of the nicotine photographs causes the nicotine-related memories to become activated and therefore, labile for interference, as previously has been shown (Dudai, 2004 ).

V. EXPERIMENTAL PROCEDURES

After screening of the participants while taking into account the inclusion and exclusion criteria (described above), they will be divided into experimental groups having similar levels of nicotine addiction and demographic background. At selected time afterwards, participants will be introduced to the TMS treatment protocol. They will be asked to refrain from smoking nicotine for two hours prior to attending the daily treatment session. Prior to stimulation onset, the participants will be presented with 'nicotine' photographs. Immediately after the offset of the photographs presentation (while memory is reactivated) the participants will be applied with real or sham rTMS stimulation. The stimulation site will be the PFC using the H-ADD coil.

Time Table:

There will be daily treatments for two weeks accompanied with assessment of the level of nicotine addiction on selected days using the above-mentioned tools. Thereafter, subjects will continue to have maintenance rTMS/sham stimulation treatment: 3 times a week for one week, two times a week in the forth and fifth week, once a week in the sixth and seventh week (see also table 2). After maintenance, participants will continue with follow up visits that will occur once a month for six months (see table 3). This protocol will allow evaluation of the short and long-term effects of the rTMS treatment with the possible fluctuations over time.

TMS procedure:

The investigators will use a Magstim Super Rapid stimulator, which produces a biphasic pulse, and our special customized equipment and coils for deep brain stimulation (Zangen, 2005 ). The TMS coils, which will be used in this study will be specific versions of the H-coil, depending on the region of stimulation. The H-coil versions used in this study, the H-ADD coil, have been tested in healthy volunteers and found to be safe and to induce some short-lasting (1 hour) cognitive alterations (Levkovitz et al., 2007, accepted). The theoretical considerations and design principles of the H-coils are explained in a previous study (Roth, 2002 ). In short, the H-ADD coil is designed to generate summation of the electric field in a specific brain region by locating coil elements at different locations around this region, all of which have a common current component which induce electric field in the desired direction .In addition, since a radial component has a dramatic effect on electric field magnitude and on the rate of decay of the electric field with distance, the overall length of coil elements which are nontangential to the skull should be minimized, and these elements as well as coil elements having current component in the opposite direction should be located as distant as possible from the brain region to be activated.

The H-ADD coil is placed on the scalp over the left motor cortex. The center of the coil is placed on the scalp with the handle pointing backward and laterally at a 45° angle away from the midline. Thus the current induced in the neural tissue is directed approximately perpendicular to the line of the central sulcus and therefore optimal for activating the corticospinal pathways transsynaptically (Kaneko et al., 1996). With a slightly suprathreshold stimulus intensity, the stimulating H-ADD coil is moved over the left hemisphere to determine the optimal position for eliciting MEPs of maximal amplitudes (the 'hot spot'). The optimal position of the coil is then marked relative to the 'hot spot' to ensure coil placement throughout the experiment. Resting motor threshold is determined to the nearest 1% of the maximum stimulator output and is defined as the minimal stimulus intensity required to produce MEPs of >50 µV in ≥5 of 10 consecutive trials at least 5 sec apart. The H-ADD coil is held in a stable coil holder ,which can be adjusted at different points relative to the 'hot spot' on the scalp.

Stimulation Protocols:

The investigators will use either sham or real H-ADD coils, which both produce similar noise and share a similar shape (as the investigators have been using in our study on healthy volunteers). Stimulation intensity will be 120% relative to the motor threshold in the 'hot spot'. PFC location will be determined as follows: 6 cm anterior to the motor 'hot spot' and symmetric.

High frequency stimulation will by applied in order to achieve activation of the stimulated brain area and possibly induce LTP like plasticity. The stimulation protocol will be 33 trains of 10 Hz for 3 seconds, ITI of 20 seconds. The total treatment duration will be 759 seconds with 990 pulses. . For that purpose the investigators have designed a special cooling system for our coils and used them successfully in our healthy volunteers study (Levkovitz et al., 2007, accepted).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, Aged 21-70 years.
* Subjects who smoke >20 cigarettes per day.
* Subjects are diagnosed as suffering from COPD
* Patients who are motivated to quit smoking.
* Patients who failed to respond to all 3 of the following anti-smoking treatments:

  1. po Bupropion (Zyban/Wellbutrin) or Varenicline (Champix)
  2. Nicotine patch/ nicotine gum
  3. CBT (Cognitive behavioral therapy)

Exclusion Criteria:

* History of a primary major psychiatric or cognitive disorder according to DSM IV.
* Current alcohol or other substance abuse or dependence.
* Alcohol or other substance abuse or dependence during the last 12 months before recruitment.
* History of or evidence of significant brain malformation or neoplasm, head injury, cerebral vascular events, neurodegenerative disorder affecting the brain or prior brain surgery.
* No neurological co-morbidity.
* No psychiatric co-morbidity.
* No psychotropic medications.
* Severe somatic co morbidity.
* Cardiac pace makers, other electronic implants, intracranial metallic particles.
* History of seizures or epileptiform activity.
* Pregnancy and lactation.
* Patients who cannot communicate reliably with the investigator or who are not likely to cope with the requirements of the experiment.
* Patients unwilling or unable to give written informed consent.
* Patients with a high risk for severe violence or suicidality as assessed during the screening interview.
* Participation in a clinical trial within the last 30 days before the beginning of this clinical trial or similar participation in another clinical trial.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-10; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Nicotine consumption(number of cigarets per day and cotinine levels )and craving (questionaires)at end of treatment (3rd week) | 3 weeks of treatment (and additional 34 weeks of maintenance & follow-up)

SECONDARY OUTCOMES:
Nicotine consumption(number of cigarets per day and cotinine levels )and craving (questionaires)at end of maintenance & follow-up(37th week) | 37 weeks (follow up)

CONTACTS AND LOCATIONS:
Overall Officials: Oded Rosenberg, M.D., Study Director — Beer Yaakov MHI; Limor Dinur Klein, Study Director — Beer Yaakov MHI
Locations (1):
- Beer-Yaacov MHC, Beer-Yaacov, Ezor Hashfela, Israel

REFERENCES:
- [Derived] Dinur-Klein L, Dannon P, Hadar A, Rosenberg O, Roth Y, Kotler M, Zangen A. Smoking cessation induced by deep repetitive transcranial magnetic stimulation of the prefrontal and insular cortices: a prospective, randomized controlled trial. Biol Psychiatry. 2014 Nov 1;76(9):742-9. doi: 10.1016/j.biopsych.2014.05.020. Epub 2014 Jun 5. PMID 25038985